CLINICAL TRIAL: NCT02286947
Title: An Open-Label, Multi-Center Study to Evaluate the Safety and Tolerability of Eteplirsen in Patients With Advanced Stage Duchenne Muscular Dystrophy
Brief Title: Safety Study of Eteplirsen to Treat Advanced Stage Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4658-204
Record Dates: First submitted 2014-10-30; First posted 2014-11-10 (Estimated); Results first posted 2019-02-20 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Muscular Dystrophy, Duchenne
Keywords: DMD; exon 51; dystrophin; dystrophy; eteplirsen; Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — eteplirsen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eteplirsen 30 mg/kg (Experimental): Participants will receive eteplirsen 30 mg/kg/week intravenous (IV) infusions, weekly, for up to 96 weeks.
  Interventions: Drug: Eteplirsen

INTERVENTIONS:
Drug: Eteplirsen — Eteplirsen solution for IV infusion
  Other Names: AVI-4658; EXONDYS 51®

SUMMARY:
The primary objective of this study is to explore safety and tolerability of eteplirsen in participants with advanced stage Duchenne muscular dystrophy (DMD) who are amenable to exon 51 skipping.

DETAILED DESCRIPTION:
This is an open-label, multi-center study to explore the safety and tolerability of eteplirsen injection in participants with advanced stage DMD with confirmed genetic mutations amenable to treatment by exon 51 skipping.

Participants will be evaluated for inclusion during a Screening/Baseline period of up to 4 weeks. Eligible participants will receive once weekly intravenous (IV) infusions of 30 mg/kg eteplirsen for 96 weeks, followed by a safety extension (not to exceed 48 weeks).

Safety will be regularly assessed throughout the study via the collection of adverse events (AEs), laboratory tests, electrocardiograms (ECGs), echocardiograms (ECHOs), vital signs, and physical examinations.

ELIGIBILITY:
Inclusion Criteria:

* Male 7 - 21 years of age
* Diagnosis of DMD with a mutation that is amenable to exon 51 skipping, confirmed by a genetic report
* Stable dose of oral corticosteroids for at least 24 weeks or has not received corticosteroids for at least 24 weeks
* Non-ambulatory, or incapable of walking ≥300 meters on the 6-Minute Walk Test (6MWT).
* Score of ≤4 on the Brooke Score for Arms and Shoulders.
* Stable cardiac and pulmonary function
* Use of contraceptives for sexually active males throughout the study
* Willing to provide consent and comply with the study

Exclusion Criteria:

* Use of any pharmacologic treatment (other than corticosteroids) within 12 weeks that may have an effect on muscle strength or function (e.g., growth hormone, anabolic steroids).
* Previous treatment with SMT C1100/BMN 195 at any time.
* Previous treatment with drisapersen (PRO051) within the last 6 months.
* Participation in any other DMD interventional clinical study within 12 weeks
* Major change in physiotherapy regimen within the past 3 months
* Major surgery within 3 months
* Presence of other clinically significant illness
* Use of an aminoglycoside antibiotic within 12 weeks or the need for this antibiotic or statin during study
* Forced vital capacity % predicted [FVC % predicted] <40%, or requiring daytime ventilation.
* Require antiarrhythmic and/or antidiuretic therapy for heart failure.
* Have a left ventricular ejection fraction (LVEF) of <40%.
* Prior or ongoing medical condition that could adversely affect the safety of the patient, make it unlikely that the course of treatment would be completed, or impair the assessment of study results.

Ages: 7 Years to 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-04-21 (Actual); Study Completion 2018-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (9):
- United States (9):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - University of California, Davis Medical Center, Sacramento, California
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - St. Louis Children's Hospital, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Seattle Children's Hospital, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted at 9 sites in the United States from November 2014 to March 2018.
Groups:
- Eteplirsen 30 mg/kg: Participants received eteplirsen 30 mg/kg intravenous (IV) infusions, once weekly, for 96 weeks.
Period: Overall Study
Arm/Group | Eteplirsen 30 mg/kg
Started | 24
Completed | 22
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all enrolled participants who received at least 1 dose of eteplirsen.
Groups:
- Eteplirsen 30 mg/kg: Participants received eteplirsen 30 mg/kg IV infusions, weekly, for 96 weeks.
Arm/Group | Eteplirsen 30 mg/kg
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.9 (3.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a participant that did not necessarily have a causal relationship with the study drug. A serious adverse event (SAE) was an AE resulting in any of the following outcomes: death; Life-threatening event; Required or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs were events that developed or worsened during the on-treatment period (defined as time from first dose of study drug and up to 28 days after last dose of study drug (up to 100 weeks) that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: From first dose of drug up to 100 weeks
Population: Analysis was performed on safety population included all participants who received at least 1 dose of eteplirsen.
Measure: Count of Participants; unit: Participants
Arm/Group | Eteplirsen 30 mg/kg
Number analyzed (Participants) | 24
Participants | 24

2. Secondary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities
Description: Laboratory parameters included hematology, clinical chemistry, urinalysis and coagulation. Data is only reported for parameters in which at least 1 participant had potentially clinically significant abnormal findings.
  Incr=increase; LLN=lower limit of normal; ULN=upper limit of normal; GGT=gamma glutamyl transferase
Time Frame: Baseline up to 100 weeks
Population: Analysis was performed on safety population included all participants who received at least 1 dose of eteplirsen.
Measure: Count of Participants; unit: Participants
Arm/Group | Eteplirsen 30 mg/kg
Number analyzed (Participants) | 24
Participants
  Sodium: Decrease of 8 or more | 3
  Sodium: Increase of 8 or more | 3
  Potassium: Decrease of 1.1 or more | 2
  Potassium: Increase of 1.0 or more | 2
  Potassium: Value > 5.5 or < 3.0 | 1
  Calcium: Decrease of 0.30 or more | 1
  Glucose: Decrease of 3.1 or more | 1
  Glucose: Increase of 3.2 or more | 6
  Albumin: Value < LLN or > ULN | 4
  Bilirubin: Incr of 10 or more | 1
  Bilirubin: Value > 1.5 x ULN | 1
  Alanine Aminotransferase: Value >= 2 x Baseline | 1
  GGT: value > 3*Baseline or > ULN | 2
  Lactate Dehydrogenase: Value >= 2 x Baseline | 1
  Creatine Kinase: Value >= 2 x Baseline | 5
  Hemoglobin: Value < LLN | 5
  Hematocrit: Value < LLN | 7
  Red Blood Cell: Value < LLN | 4
  White Blood Cell: Value < LLN or > 1.5 x ULN | 5
  Platelets: Value < 150 or < 200 | 1
  Neutrophils: Value > 1.5 x ULN or < 1000 | 7
  Lymphocytes: Value < LLN | 6
  Monocytes: Value < LLN | 14
  Eosinophils: Value > 1.5 x ULN or < LLN | 2
  Basophils: Value < LLN or > ULN | 2
  Urine Protein: Value > 1+ | 5

3. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities in Vital Signs
Description: Vital sign parameters included systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR), and body temperature. Data is only reported for parameters in which at least 1 participant had potentially clinically significant abnormal vital sign findings.
Time Frame: Baseline up to 100 weeks
Population: Analysis was performed on safety population included all participants who received at least 1 dose of eteplirsen.
Measure: Count of Participants; unit: Participants
Arm/Group | Eteplirsen 30 mg/kg
Number analyzed (Participants) | 24
Participants
  DBP: Less than 40 mmHG | 1
  DBP: Greater than 90 mmHg | 12
  SBP: Less than 80 mmHg | 4
  SBP: Greater than 130 mmHG | 17
  HR: Less than 50 beats per minute (bpm) | 1
  HR: Greater than 130 bpm | 15

4. Secondary Outcome: Number of Participants With at Least One Potentially Clinically Significant Abnormalities in Physical Examinations
Description: Physical examinations, full and brief, were performed by the Investigator, a physician Sub-Investigator, or a Nurse Practitioner (if licensed in the state or province to perform physical examinations). Full physical examinations included examination of general appearance; head, ears, eyes, nose, and throat; heart; lungs; chest; abdomen; skin; lymph nodes; and musculoskeletal and neurological systems. Brief physical examinations included examination of general appearance; head, ears, eyes, nose, and throat; heart; lungs; chest; abdomen; and skin.
Time Frame: Baseline up to 100 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Eteplirsen 30 mg/kg
Number analyzed (Participants) | 24
Participants | 23

5. Secondary Outcome: Number of Participants With Abnormalities in Electrocardiograms (ECGs)
Description: Twelve-lead ECGs and Holter ECGs were performed at a consistent time of day throughout the study. Electrocardiograms were performed only after the patient was in the supine position, resting, and quiet for a minimum of 15 minutes. The ECG was manually reviewed and interpreted by medically qualified personnel using a central vendor according to prespecified criteria. The Investigator reviewed the results of the centrally read ECG report and determined if the findings were clinically significant. Data is only reported for parameters in which at least 1 participant had potentially clinically significant abnormal ECG findings.
  msec=milliseconds; QTcF=QT interval corrected with Fridericia's method
Time Frame: Baseline up to 100 weeks
Population: Analysis was performed on safety population included all participants who received at least 1 dose of eteplirsen.
Measure: Count of Participants; unit: Participants
Groups:
- Eteplirsen 30 mg/kg: Participants received eteplirsen 30 mg/kg intravenous (IV) infusions, weekly, for 96 weeks.
Arm/Group | Eteplirsen 30 mg/kg
Number analyzed (Participants) | 24
Participants
  Heart Rate: >120 beats/minute | 6
  QTcF: Increase of 60 or more msec | 1

6. Secondary Outcome: Number of Participants With Abnormalities in Echocardiograms (ECHO)
Description: Standard, 2-dimensional ECHOs were performed at a consistent time of day throughout the study. The ECHO was reviewed and interpreted by medically qualified personnel using a central vendor according to prespecified criteria. Ejection fraction was noted. The Investigator reviewed the results of the ECHO report and determined if the findings were clinically significant.
  LEVF=left ventricular ejection fraction
Time Frame: Baseline up to 100 weeks
Population: Analysis was performed on safety population included all participants who received at least 1 dose of eteplirsen.
Measure: Count of Participants; unit: Participants
Arm/Group | Eteplirsen 30 mg/kg
Number analyzed (Participants) | 24
Participants
  LEVF: <55% | 0
  Fractional Shortening: <28% | 6

ADVERSE EVENTS:
Time Frame: Baseline up to Week 100
Arm/Group | Eteplirsen 30 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 4/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eteplirsen 30 mg/kg (N=24)
Extremity contracture (Musculoskeletal and connective tissue disorders) | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eteplirsen 30 mg/kg (N=24)
Nasopharyngitis (Infections and infestations) | 14
Upper respiratory tract infection (Infections and infestations) | 6
Ear infection (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 3
Pharyngitis streptococcal (Infections and infestations) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2
Contusion (Injury, poisoning and procedural complications) | 6
Procedural pain (Injury, poisoning and procedural complications) | 4
Joint injury (Injury, poisoning and procedural complications) | 3
Ligament sprain (Injury, poisoning and procedural complications) | 3
Foot fracture (Injury, poisoning and procedural complications) | 2
Skin abrasion (Injury, poisoning and procedural complications) | 2
Soft tissue injury (Injury, poisoning and procedural complications) | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2
Vomiting (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 4
Abdominal discomfort (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 8
Acne (Skin and subcutaneous tissue disorders) | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 2
Rash papular (Skin and subcutaneous tissue disorders) | 2
Catheter site pain (General disorders) | 5
Infusion site bruising (General disorders) | 4
Catheter site bruise (General disorders) | 3
Pyrexia (General disorders) | 3
Chest pain (General disorders) | 2
Infusion site pain (General disorders) | 2
Headache (Nervous system disorders) | 8
Dizziness (Nervous system disorders) | 2
Breath sounds abnormal (Investigations) | 3
Protein urine present (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Depression (Psychiatric disorders) | 2
Renal pain (Renal and urinary disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The most restrictive relevant agreement provides that the PI can only publish the study results with the approval of Sponsor.

DOCUMENTS (2):
  • Study Protocol (2016-07-05): https://cdn.clinicaltrials.gov/large-docs/47/NCT02286947/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT02286947/SAP_001.pdf